CLINICAL TRIAL: NCT03042715
Title: Psychological Intervention to Promote Coping for Caregivers of Patients Undergoing Hematopoietic Stem Cell Transplantation (HCT)
Brief Title: Psychological Intervention for Caregivers of Patients Undergoing Hematopoietic Stem Cell Transplantation (HCT)
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Areej El-Jawahri, MD, Massachusetts General Hospital
Other Study IDs: 16-522
Record Dates: First submitted 2017-01-28; First posted 2017-02-03 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Stem Cell Transplant Complications
Keywords: Supportive Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Psychological Intervention refinement: * Eight weekly sessions in-person or via telephone
  * Qualitative interviews
  * Feedback from 5-10 caregivers to refine the intervention.
  Interventions: Behavioral: Qualitative Interviews

INTERVENTIONS:
Behavioral: Qualitative Interviews — phase 1 of the study entail refining the psychological intervention based on caregivers' feedback

SUMMARY:
This research study is evaluating a psychological intervention for caregivers of patients undergoing stem cell transplantation.

Phase 1 will include a qualitative phase to refine the intervention to specifically target the needs of caregivers

Phase 2 of the trial will transition to an interventional randomization clinical trial

DETAILED DESCRIPTION:
The purpose of this study is to find out whether a psychological intervention can help caregivers learn effective coping methods during their loved one's transplant process and make the experience of being a caregiver more manageable.

Phase 1 of the project entails using qualitative interviews with caregivers to further refine the intervention. The psychological intervention will take place over the course of a patient transplant in a series of eight sessions. A trained behavioral psychologist will meet with the participant or talk with them over the telephone for 30-45 minutes at a time to discuss the caregiver experience and to help develop effective skills to support the patient as well as the participant over the course of the transplant.

Upon the completion of the sessions, the investigators will have a short, audio-recorded exit interview to obtain the participant's feedback on the intervention. At the participant's convenience, this interview will be conducted in-person or over the phone. The investigators will use the feedback to improve the intervention before further testing its efficacy in phase 2, a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregivers (≥18 years) of patients undergoing HCT at MGH.
* A relative or a friend who either lives with the patient or has in-person contact with him or her at least twice per week and is identified as the primary caregiver for transplant
* Ability to speak English or able to complete questionnaires with minimum assistance of an interpreter.

Exclusion Criteria:

* Significant uncontrolled psychiatric disorder (psychotic disorder, bipolar disorder, major depression)
* Other co-morbid disease (dementia, cognitive impairment), which the treating clinician believes prohibits the ability to participate in study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers will be recruited during the patient transplant consent visit, which typically occurs 2-4 weeks prior to admission for HCT. Caregivers are required to attend the HCT consent visit with the patient.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Qualitative Refinement: this clinical trials.gov report is focused on the qualitative refinement phase of the project.
Period: Overall Study
Arm/Group | Qualitative Refinement
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Psychological Intervention Refinement: * Eight weekly sessions in-person or via telephone
  * Qualitative interviews
  * Feedback from 5-10 caregivers to refine the intervention.
  Qualitative Interviews: phase 1 of the study entail refining the psychological intervention based on caregivers' feedback
Arm/Group | Psychological Intervention Refinement
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 4
  male | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pilot Qualitative Refinement of the Caregiver Intervention
Description: qualitative data to develop and refine the caregiver intervention
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Qualitative Refinement: pilot qualitative refinement of intervention
Arm/Group | Qualitative Refinement
Number analyzed (Participants) | 6
Participants
  intervention length is feasible | 5
  session length is appropriate | 5
  preferred fewer visits | 3
  focus on mindfulness is appropriate | 5

ADVERSE EVENTS:
Time Frame: qualitative refinement of an intervention, no adverse events reported during the entire study period (1 year). all caregivers were followed for a total of 3 months during the intervention refinement
Arm/Group | Qualitative Refinement
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT03042715/Prot_SAP_000.pdf